CLINICAL TRIAL: NCT06763250
Title: Risk Factors Influencing Textbook Outcomes in PD Surgery-a Single-center Analysis
Brief Title: In This Study, a Retrospective Analysis Was Conducted to Explore the Risk Factors for Patients Undergoing Pancreaticoduodenal Surgery (PD) to Achieve TO, and a Nomogram Prediction Model Was Further Established to Promote the Standardization and Standardization of PD Surgical Quality Evaluation.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: luokai zhang (Other)
Responsible Party: Sponsor-Investigator, luokai zhang, Changzhou Second People's Hospital, Jiangsu Province, Changzhou No.2 People's Hospital
Organization: Changzhou No.2 People's Hospital (Other)
Other Study IDs: CN CZEY
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Carcinoma; Cholangiocarcinoma; Pancreaticoduodenectomy
Keywords: textbook outcome; pancreatic carcinoma; cholangiocarcinoma; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- We divided the clinical data into a TO group and a non-TO group through retrospective analysis: A textbook outcome (TO) of pancreatic surgery based on an international expert consensus, No postoperative hemorrhage of grade B/C, no postoperative pancreatic fistula of grade B/C, no biliary leakage of grade B/C, Clavien-Dindo complication grade < Ⅲ, no death during hospitalization or within 30 days after surgery, and no re-admission within 30 days after discharge were integrated as a comprehensive index. It can reflect the ideal surgical outcome. We divided the clinical data into a TO group and a non-TO group through retrospective analysis. In order to promote the standardization and standardization of PD surgical quality assessment.

SUMMARY:
This study is committed TO exploring the risk factors affecting patients receiving pancreaticoduodenal surgery (PD) to achieve TO by retrospective analysis of clinical data of patients receiving PD surgery in Changzhou Second People Hospital from January 2016 to December 2024, and further establishing a nomogram prediction model. In order to promote the standardization and standardization of PD surgical quality assessment.

DETAILED DESCRIPTION:
As we all know, pancreaticoduodenectomy (whipple) involving multiple organ reconstruction for pancreatic cancer is known as the "surgical ceiling", but because of its high postoperative complication rate and poor prognosis, a standardized surgical quality assessment system covering the whole perioperative period is urgently needed. The concept of the textbook ending was born.it first appeared in a 2013 study by Kolfschoten et al for colorectal cancer, in which textbook outcomes were evaluated in an all or none ,manner against six independent expected outcome measures: There were no deaths in hospital or within 30 days after surgery, radical resection, no re-intervention, no stomy, no serious postoperative complications, and no prolonged hospital stay. That is, when patients meet the above six indicators at the same time, they are defined as achieving a textbook outcome .In our study, the textbook outcome is the primary outcome, and the reverse is the secondary outcome.This study is committed TO exploring the risk factors affecting patients receiving pancreaticoduodenal surgery (PD) to achieve TO by retrospective analysis of clinical data of patients receiving PD surgery in Changzhou Second People Hospital from January 2016 to December 2024, and further establishing a nomogram prediction model. In order to promote the standardization and standardization of PD surgical quality assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received radical PD surgery and whose pathological findings were clear tumors;
2. Complete clinical data preservation.

Exclusion Criteria:

1. Palliative resection; 2. Tumor metastasis or other primary tumors; 3. Combined with severe organ dysfunction; 4. Postoperative pathology was not clear tumor.

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From the 260 specimens collected so far in this study, we obtained the description of the study population. In terms of age, 6.53% of the samples were less than 50 years old, 13.84% were more than or equal to 50 years old and 60 years old, 46.54% were more than or equal to 60 years old and 70 years old, 29.23% were more than or equal to 70 years old and 3.86% were more than or equal to 80 years old. In terms of gender, 57.31% of the sample were male and 42.69% were female. All the samples in this study were Han. 98.85% of the sample were married. The population samples for this study were all from the Second People's Hospital of Changzhou City.The risk factors affecting the textbook outcome of PD surgery in this study population were: 1. Diabetes; 2. Preoperative bile duct inflammation; 3. Intraoperative pancreatic duct diameter; 4; Vascular invasion; 5. Duration of operation; 6. Surgical method.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Achieve TO as the main ending | from January 2016 to August 2024
  We expected TO collect 280 PD surgery patients, 262 cases have been collected, of which 158 cases achieved TO as the main outcome, the TO rate is 60.31%.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Changzhou, Jiangsu Province, China, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma L, Wu S, Cheng Y, Gao Y, Fan J, Zhu C. Laparoscopic duodenum-preserving total pancreatic head resection for benign and low-grade malignant tumors close to the accessory papilla (a case series). Surg Endosc. 2025 Oct 23. doi: 10.1007/s00464-025-12236-9. Online ahead of print. PMID 41128852